CLINICAL TRIAL: NCT05411614
Title: A Randomised Controlled Trial Comparing Convergent Hybrid Ablation to Catheter Ablation in Patients With Persistent Atrial Fibrillation and Heart Failure
Brief Title: Hybrid Ablation of Atrial Fibrillation in Heart Failure
Acronym: HALT AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. George's Hospital, London (Other)
Responsible Party: Principal Investigator, Riyaz Kaba, Consultant in Cardiology and Cardiac Electropysiology, St. George's Hospital, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021.0137
Record Dates: First submitted 2022-05-20; First posted 2022-06-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Persistent Atrial Fibrillation; Atrial Fibrillation, Persistent; Atrial Arrhythmia; Atrial Fibrillation; Heart Failure; Left Ventricular (LV) Systolic Dysfunction
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Clinical study. 1:1 randomised. Convergent Hybrid Ablation Procedure versus standalone endocardial catheter ablation).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convergent Hybrid Ablation +/- Left Atrial Appendage Exclusion (Experimental): Staged Convergent Hybrid Ablation Procedure
  Stage 1 - Minimally-Invasive Surgical Epicardial Ablation Procedure +/- concomitant LAA exclusion.
  Stage 2 - Endocardial Catheter Ablation
  Interventions: Device: AtriCure EPi-Sense-AF Guided Coagulation System +/- Atriclip; Device: Endocardial Catheter Ablation
- Standard Endocardial Catheter Ablation (Active Comparator): Standard endocardial catheter ablation
  Interventions: Device: Endocardial Catheter Ablation

INTERVENTIONS:
Device: AtriCure EPi-Sense-AF Guided Coagulation System +/- Atriclip — Minimally-invasive epicardial ablation +/- left atrial appendage exclusion using an epicardial clip, combined with endocardial radiofrequency catheter ablation
  Other Names: Convergent Hybrid Epicardial Endocardial Ablation plus/minus left atrial appendage exclusion
  Arms: Convergent Hybrid Ablation +/- Left Atrial Appendage Exclusion
Device: Endocardial Catheter Ablation — Standard percutaneous endocardial catheter ablation of atrial fibrillation
  Other Names: Percutaneous Catheter Ablation

SUMMARY:
A randomised controlled trial to assess the efficacy of staged hybrid ablation when compared with standard catheter ablation in patients with non-paroxysmal atrial fibrillation (AF) and Heart Failure

DETAILED DESCRIPTION:
The objective of this randomized study is to evaluate the safety and efficacy of Convergent hybrid ablation when compared to standard catheter ablation in patients with non-paroxysmal AF and heart failure.

Patients will be randomised in a 1:1 ratio. The primary efficacy endpoint will be freedom from persistent atrial arrhythmia (measured from the end of a 3-month blanking period up to 24 months (12 and 24 months).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Persistent or Long-standing Persistent AF
* Dilated left atrium (at least moderately dilated)
* Suitable for either procedure
* LVEF < 50%

Exclusion Criteria:

* Not yet optimised from a medical or lifestyle perspective for AF or heart failure
* Unable to provide written consent
* Previous open-heart surgery
* Active infection, oesophageal ulcer stricture or oesophageal varices
* Prior catheter ablation of atrial fibrillation (prior ablation for atrial flutter / supraventricular tachycardia or ventricular arrhythmia acceptable)
* Contraindication to anticoagulation, or active thrombus in the left atrium despite therapeutic anticoagulation
* Severe valvular heart disease
* Unstable coronary artery disease
* Uncontrolled ventricular arrhythmia
* Heart attack or stroke within the last 90 days
* Pregnant, breastfeeding, or women of childbearing age who plan to get pregnant within six months
* Severe concomitant condition or presence of an implanted device that would preclude the patient from undergoing trial procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from persistent atrial arrhythmia after a single procedure (either the completed hybrid ablation or catheter ablation) off Class I or III medications | Measured from the end of a 3-month blanking period at 12 and 24 months
  Recurrence of persistent atrial arrhythmia during follow-up months).

SECONDARY OUTCOMES:
Safety Endpoint | Measured as early (within 30- days) and late (> 30 days) after each procedure or part of procedure
  Safety endpoint of severe and non-severe complications as defined in the protocol
Freedom from any atrial arrhythmia lasting > 30 seconds after a single completed procedure on class I/III medications | Measured from the end of a 3- month blanking period at 12 and 24 months
  Recurrence of any atrial arrhythmia > 30 seconds on or off class I / III medications, considering any repeat ablation procedures
Freedom from atrial arrhythmias after any redo procedures (on or off class I or III medications) | Measured from the end of a 3- month blanking period at 12 and 24 months
  Recurrence of any atrial arrhythmia > 30 seconds on or off class I / III medications, considering any repeat ablation procedures
To assess left ventricular structural remodelling and change in ventricular function in response to either procedure | Pre-procedure and at 12 and 24 months post-procedure
  Left ventricular ejection fraction as recorded on transthoracic echocardiography (TTE)
To assess left atrial remodelling in response to either technique. | Pre-procedure and up to 12 and 24 months post-procedure
  Left atrial dimensions/function on Echocardiography
To evaluate the effects of the interventions on the patient's symptoms and quality of life (EHRA Score) | Pre-procedure and at 12 and 24 months post-procedure
  Change in European Heart Rhythm Association (EHRA) AF Symptom score
To evaluate the effects of the interventions on the patient's symptoms and quality of life (NYHA Class). | Pre-procedure and at 12 and 24 months post-procedure
  Change in New York Heart Association (NYHA) class
To evaluate the effects of the interventions on the patient's quality of life (EQ5D) | Pre-procedure and at 12 and 24 months post-procedure
  Change in EuroQol Quality of life Score (EQ5D)
To evaluate the effects of the interventions on the patient's quality of life (AFEQT) | Pre-procedure and at 12 and 24 months post-procedure
  Change in Atrial Fibrillation Effect on Quality of Life Score (AFEQT)

CONTACTS AND LOCATIONS:
Overall Officials: Riyaz A Kaba, Principal Investigator — St Georges Hospital NHS Trust; Omar Ahmed, Principal Investigator — St Georges Hospital NHS Trust
Locations (7):
- United Kingdom (7):
  - Ashford & St Peters Hospital NHS Trust, Chertsey
  - Epsom General Hospital, Epsom
  - Cromwell Hospital, London
  - Royal Surrey County Hospital, London
  - St Anthonys Hospital, London
  - St Georges at Kingston Hospital, London
  - St Georges University of London, London

IPD SHARING:
Plan to Share IPD: No